CLINICAL TRIAL: NCT02503436
Title: C-PATROL - a Single Arm, Prospective Non-interventional Study (NIS) to Collect Clinical and Patient Reported Outcome Data in an Olaparib Treated BRCAm+ PSR Ovarian Cancer Population
Brief Title: C-PATROL - Non-interventional Study (NIS) to Collect Clinical and Patient Reported Outcome Data in an Olaparib Treated BRCAm+ PSR Ovarian Cancer Population
Acronym: C-PATROL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0816R00009
Record Dates: First submitted 2015-07-08; First posted 2015-07-21 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Ovarian Cancer, Hereditary Ovarian Cancer Syndrome
Keywords: Ovarian Cancer, Fallopian Tube Cancer, primary peritoneal cancer, BRCA1 Gene, BRCA2 Gene
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Fanconi Anemia, Complementation Group D1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 84 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of the proposed non-interventional study is to obtain real-world effectiveness, safety and treatment patterns data of patients with BRCAm+ (Breast Cancer Gene(s) mutation positive) platinum sensitive relapsed (PSR) ovarian cancer in German hospitals and outpatient practices treated with olaparib.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Women aged ≥ 18 years
* Patients with platinum sensitive relapsed high grade epithelial ovarian cancers (including primary peritoneal and/or fallopian tube cancer). (Platinum sensitive disease is defined as disease progression ≥6 months after completion of their last dose of platinum based chemotherapy. Patients must be currently in response to platinum-based chemotherapy. For the last chemotherapy course immediately prior to enrolment on the study, patients must be, in the opinion of the investigator, in response (partial or complete), following completion of this chemotherapy course.
* Documented BRCA mutations (germline and/or somatic mutation in BRCA1 (Breast Cancer gene 1) and/or BRCA2 (Breast Cancer gene 2) that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function))
* Patients should be in line with the specifications mentioned in the German LYNPARZA (olaparib) SmPC (Summary Product Characteristics) for hard capsules or tablets.
* Patients are able to read and understand German, English, Turkish or Arabic

Exclusion Criteria:

* Known hypersensitivity to olaparib or any of the excipients of the drug
* Patients who have started olaparib monotherapy for more than 14 days before giving their informed consent
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 patients in 80 sites (approx. 40 hospitals and 40 outpatient practices) in Germany. Each site should enrol 2-30 patients
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
To assess clinical effectiveness of olaparib maintenance monotherapy by assessment of progression free survival (PFS) in patients with BRCAm+ ovarian cancer. Methods and time intervals for tumor assessment depend on the investigator's decision. | Date of first documented dose of olaparib to the date of progression (as judged by the investigator) or death (of any cause) whichever occurred before, assessed approximately up to 84 months

SECONDARY OUTCOMES:
To collect and explore real-life data on patient outcomes in terms of Overall Survival (OS) | Date of first documented dose of olaparib to death of any cause, assessed approximately up to 84 months
Time to first subsequent therapy (TFST) | Date of first documented dose of olaparib to date of first administration of first subsequent therapy or death if this occurs before commencement of first subsequent treatment, assessed approximately up to 84 months
Progression-free survival 2 (PFS2) | Date of first administration of first subsequent therapy to date of progression as assessed by the investigator or death, assessed approximately up to 84 months
Time to second subsequent therapy (TSST) | Date of first documented dose of olaparib to date of first administration of second subsequent therapy or death if this occurs before commencement of second subsequent treatment, assessed approximately up to 84 months
Time to discontinuation of olaparib monotherapy (TDO) | Date of first documented dose of olaparib montherapy to date of last documented dose of olaparib monotherapy or death whichever occurred before, assessed approximately up to 84 months
Assessment of health-related quality of life (HRQoL) in patients participating in the study. | Date of first visit to last visit. HRQoL are collected every 3 months up to 84 months
  Health related quality of life (HRQoL): Assessment of general cancer-associated and specific ovarian cancer associated parameters by use of standardized HRQoL questionnaires:
  * Functional assessment of Cancer Therapy for Patients with Ovarian Cancer (FACT-O)
  * Functional Assessment of Chronic Illness - Fatigue (FACIT-Fatigue)
  * Functional Living Index - Emesis (FLIE)
Safety of Olaparib: collection of Adverse Events (AE) | Date of first documented dose of Olaparib to last visit, assessed approximately up to 84 months
  Type and frequeny of adverse event (AE), intensity, causal relationship to olaparib, outcome, seriousness, management of adverse event

CONTACTS AND LOCATIONS:
Locations (68):
- Germany (68):
  - Research Site, Amberg
  - Research Site, Aschaffenburg
  - Research Site, Augsburg
  - Research Site, Bad Homburg
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Bottrop
  - Research Site, Brandenburg
  - Research Site, Braunschweig
  - Research Site, Bremen
  - Research Site, Chemnitz
  - Research Site, Coburg
  - Research Site, Cologne
  - Research Site, Donauwörth
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Eutin
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Fürstenwalde
  - Research Site, Georgsmarienhütte
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Heidenheim
  - Research Site, Hildesheim
  - Research Site, Homburg/Saar
  - Research Site, Jena
  - Research Site, Karlsruhe
  - Research Site, Kassel
  - Research Site, Kempten
  - Research Site, Kiel
  - Research Site, Krefeld
  - Research Site, Kulmbach
  - Research Site, Landshut
  - Research Site, Lübeck
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, Mönchengladbach
  - Research Site, Mutlangen
  - Research Site, München
  - Research Site, Münster
  - Research Site, Nuremberg
  - Research Site, Oberhausen
  - Research Site, Osnabrück
  - Research Site, Paderborn
  - Research Site, Plauen
  - Research Site, Regensburg
  - Research Site, Rosenheim
  - Research Site, Rostock
  - Research Site, Saarbrücken
  - Research Site, Schwerin
  - Research Site, Singen
  - Research Site, Solingen
  - Research Site, Stralsund
  - Research Site, Stuttgart
  - Research Site, Traunstein
  - Research Site, Troisdorf
  - Research Site, Tübingen
  - Research Site, Wiesbaden
  - Research Site, Wolfsburg
  - Research Site, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816R00009&attachmentIdentifier=c164b9da-57d5-441c-a64c-cda2353493cc&fileName=D0816R00009_CSR_Synopsis.pdf&versionIdentifier=